CLINICAL TRIAL: NCT01121705
Title: Multicenter Study on Efficacy of New Therapeutic Schedules With Peg-Interferon alpha2b and Ribavirin in Patients With Genotype 3 Chronic HCV( Hepatitis C Virus) Infection
Brief Title: Efficacy Study of New Therapeutic Schedules in Naive Hepatitis C Virus (HCV) Patients Infected With Genotype 3 (HCV-3)
Acronym: genotype-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Casa Sollievo della Sofferenza IRCCS (Other)
Responsible Party: Angelo Andriulli, MD, IRCCS "Casa Sollievo della Sofferenza"
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007-00437470
Record Dates: First submitted 2010-05-04; First posted 2010-05-12 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2009-06

CONDITIONS: Chronic Hepatitis
Keywords: genotype 3; Combination treatment; Short treatment
MeSH Terms: conditions — Hepatitis, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A1. standard duration (No Intervention): Patients were randomly assigned in a 1:1 ratio to two treatment arms. In the standard treatment group (A1), patients were treated for 24 weeks irrespective of the HCV RNA status at week 4 with Peg-interferon alfa-2b at a dose of 1.5 mcg per kilogram of body weight weekly in combination with oral ribavirin administered at a dose of 1000 mg/day for patients with a weight <75 kg or 1200 mg/day for those with a weight of ≥75 kg. Patients enrolled in Arm A1 will be treated for standard 24 weeks duration of treatment with standard dosages of PegInterferon alpha 2b and weight-based dosages of ribavirin.
- B 1 I or II (Experimental): In the variable treatment group, patients with a virologic response at week 4 will receive treatment for 12 weeks and those without a virologic response at 4 weeks treatment for 36 weeks. Patients without RVR will be treated for 24 or 36 weeks and labelled (B1I) or (B1II, respectively Intervention: different durations of treatment for patients without RVR
  Interventions: Drug: Peg Interferon alpha2b + Ribavirin

INTERVENTIONS:
Drug: Peg Interferon alpha2b + Ribavirin — B 1 I or II: Experimental
  variable duration of treatment group according with RVR. In case of RVR present patients will be treated for 12 weeks. Patients without RVR will be treated for 24 (B1I) or 36 (B1II)weeks: different duration of treatment for patients without RVR
  Other Names: variable
  Arms: B 1 I or II

SUMMARY:
The study aimed at evaluating whether current 24 weeks length of combination treatment is appropriate or not for patients with HCV genotype 3 infection.

DETAILED DESCRIPTION:
Patients are randomized to standard length of treatment or to a variable duration: 12 weeks for patients with undetectable HCVRNA at week 4 or 24 or 36 weeks for those with detectable HCV RNA at week 4.

ELIGIBILITY:
Inclusion Criteria:

* Naive HCV patients
* HCVRNA positive
* Normal TSH
* ANA <1:160

Exclusion Criteria:

* Portal hypertension
* Renal failure
* HBsAg or HIV
* Alcohol consumption >30 g/day
* Active IV drug use
* Chronic systemic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2007-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Sustained virological response (SVR) | 6 months after the end of treatment
  The primary measure of efficacy will be HCV RNA not detectable in the serum 24 weeks after the end of therapy (SVR). In addition, virological response at the end of treatment and relapse rates will be calculated for each groups. Two analyses will be performed: 1) intention-to-treat analysis; 2) per-protocol analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Mangia, MD, Study Director — IRCCS - San Giovanni Rotondo
Locations (8):
- Italy (8):
  - Ospedale Civile, Sassari, Sassari
  - Ospedale Civile, Canossa
  - Ospedale Casarano, Casarano
  - IRCCS "De Bellis", Castellana Grotte
  - Ospedale "Garibaldi", Catania
  - Ospedale "S.Camillo", Rome
  - Università Cattolica Sacro Cuore Roma, Rome
  - Ospedale Venosa, Venosa

REFERENCES:
- [Background] Andriulli A, Mangia A, Iacobellis A, Ippolito A, Leandro G, Zeuzem S. Meta-analysis: the outcome of anti-viral therapy in HCV genotype 2 and genotype 3 infected patients with chronic hepatitis. Aliment Pharmacol Ther. 2008 Aug 15;28(4):397-404. doi: 10.1111/j.1365-2036.2008.03763.x. Epub 2008 Jun 11. PMID 18549461